CLINICAL TRIAL: NCT01802437
Title: An Adaptive Treatment Strategy for Adolescent Depression
Acronym: PTAD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1110M05542
Record Dates: First submitted 2013-02-01; First posted 2013-03-01 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Talk Therapy 4-Week Decision Point (Experimental): Interpersonal psychotherapy that focuses on an adolescents relationship and communication skills in the context of of their depression. After 4 weeks of therapy, participants with at less than a 20% reduction in Hamilton Rating Scale for Depression (HRSD) score will be further randomized into 2 groups, increased dose of interpersonal psychotherapy frequency or introduction of fluoxetine therapy starting with 10 mg per day for the first week and 20 mg per day in the following 5 weeks. If HRSD scores meet target, patients continue to receive initial dose of interpersonal psychotherapy
  Interventions: Drug: Fluoxetine; Behavioral: Increased Dose of Interpersonal Psychotherapy; Behavioral: Continue to Receive Initial Dose of Interpersonal Psychotherapy
- Talk Therapy 8-Week Decision Point (Experimental): Interpersonal psychotherapy that focuses on an adolescents relationship and communication skills in the context of of their depression. After 8 weeks of therapy, participants with at less than a 40% reduction in Hamilton Rating Scale for Depression (HRSD) score will be further randomized into 2 groups, increased dose of interpersonal psychotherapy or introduction of fluoxetine therapy starting with 10 mg per day for the first week and 20 mg per day in the following 5 weeks. If HRSD scores meet target, patients continue to receive initial dose of interpersonal psychotherapy.
  Interventions: Drug: Fluoxetine; Behavioral: Increased Dose of Interpersonal Psychotherapy; Behavioral: Continue to Receive Initial Dose of Interpersonal Psychotherapy

INTERVENTIONS:
Drug: Fluoxetine — If Hamilton Rating Scale for Depression scores do not meet target reductions (20% reduction for 4-week decision point or 40% reduction for 8-week decision point), adolescents will be further randomized to an increase in therapy (4 extra therapy sessions) or fluoxetine therapy. Adolescents who receive pharmacotherapy will be prescribed fluoxetine for 12 weeks. The dosage schedule will be 10 mg per day for the first week and 20 mg per day for the following 5 weeks. If no treatment response is observed by week 6, the dosage can be increased to 40 mg per day. Pharmacotherapy sessions will be scheduled weekly for the first 4 weeks and every other week thereafter. If no treatment response was observed by the sixth week, the dosage could be increased to 40 mg per day.
  Other Names: Prozac
Behavioral: Increased Dose of Interpersonal Psychotherapy — If Hamilton Rating Scale for Depression scores do not meet target reductions (20% reduction for 4-week decision point or 40% reduction for 8-week decision point), adolescents will be further randomized to an increased dose of interpersonal psychotherapy (4 extra therapy sessions) or fluoxetine.
Behavioral: Continue to Receive Initial Dose of Interpersonal Psychotherapy — If Hamilton Rating Scale for Depression scores meet target reductions (20% reduction for 4-week decision point or 40% reduction for 8-week decision point), adolescents will be assigned to continue initial dose of interpersonal psychotherapy.

SUMMARY:
The purpose of the study is:

1. to find out how long teenagers getting talk therapy (interpersonal psychotherapy) for depression should get therapy before the therapist decides whether or not the teenager is improving enough, and
2. to compare two ways of providing treatment to teenagers who have not improved enough.

DETAILED DESCRIPTION:
Study Procedures

This study has three phases:

1. The screening and eligibility phase:

   Parent and child will conduct an initial evaluation that will last about 4 hours. The evaluator will ask questions and the participant will complete forms about his/her mood and behavior. This intake appointment will determine eligibility for the study.
2. The treatment phase: The child would begin a kind of talk therapy called interpersonal psychotherapy. The goal of the therapy is to decrease teenagers' depression by helping them improve their relationships and communication skills. The child will attend 12 therapy appointments over the course of 16 weeks. Each appointment will be 50 minutes long.

   If the child is doing well with standard interpersonal therapy, it will be continued without change. If the child has not improved enough, we will change the treatment plan in one of two ways. The choice will be based on chance (sort of like flipping a coin) and will be done by a computer.

   ***Your child will attend 16 therapy appointments (that is four additional sessions). These additional four sessions will be scheduled so that your child will attend therapy twice a week for a period of four weeks.

   -OR-

   ***Your child will continue to attend 12 therapy appointments over the course of 16 weeks and your child will also be prescribed an antidepressant medication called fluoxetine. Fluoxetine is also known as Prozac. Prozac has been approved by the Food and Drug Administration for use in the treatment of depressed teenagers. You will be responsible for paying for the medication.

   At four points during the treatment phase (week 4, week 8, week 12, and week 16), parent and child will be asked to complete forms and interviews to see how the child is doing. The evaluations at weeks 4, 8, and 12 will take approximately 1 hour. At the end of treatment, parent and child will have a longer meeting with the evaluator (4 hours) to see if the treatment your child got was helpful. During these meetings, we will also ask participants to fill out some forms about your mood and mental health treatment.
3. The follow-up phase: Parent and child will be asked to return for a follow-up assessment 4 months after the child completes the treatment phase to see how he or she is doing. Parent and child will be asked to complete forms and interviews. This meeting will take approximately 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent meets DSM-IV-TR criteria for a diagnosis of Major Depressive Disorder, Dysthymia, or Depressive Disorder NOS; demonstrate symptoms of depression (CDRS-R > 35); and demonstrate impairment in general functioning (CGAS < 65).
* Adolescents and parents must be English-speaking

Exclusion Criteria:

* Adolescent meets criteria for a diagnosis of Schizophrenia, Bipolar Disorder, Psychosis, Substance Abuse, OCD, Conduct Disorder, Eating Disorder, PDD, or intellectual disability disorder.
* Depressed adolescents who are actively suicidal with a plan and/or intent
* Adolescent that are already receiving treatment for depression or if they are taking medication for a psychiatric diagnosis other than ADHD. Depressed adolescents with a comorbid diagnosis of ADHD who are on a stable dose of stimulant medication (> 3 months) will be eligible to participate in the studies.
* Adolescent that have already received an adequate trial of IPT-A or fluoxetine.
* Female adolescents who are pregnant, breastfeeding, or having unprotected sexual intercourse.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Gunlicks-Stoessel, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Department of Psychiatry, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point
Started | 20 | 20
Completed | 16 | 16
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Talk Therapy 8-Week Decision Point: Interpersonal psychotherapy that focuses on an adolescents relationship and communication skills in the context of of their depression. After 8 weeks of therapy, participants with at less than a 40% reduction in Hamilton Rating Scale for Depression (HRSD) score will be further randomized into 2 groups, increased dose of interpersonal psychotherapy or introduction of fluoxetine therapy starting with 10 mg per day for the first week and 20 mg per day in the following 5 weeks. If HRSD scores meet target, patients continue to receive initial dose of interpersonal psychotherapy.
  Interpersonal Psychotherapy: Adolescent randomized to an increase in therapy (4 extra therapy sessions)
- Total: Total of all reporting groups
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.8) | 14.8 (1.8) | 14.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 16 | 32
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Children's Depression Rating Scale-Revised Score (CDRS-R) [Mean (Standard Deviation); unit: score] — The CDRS-R is a clinician-administered semi-structured interview that assesses symptoms of depression experienced during the previous 2-weeks. The first 14 items are rated on the basis of an interview. The remaining 3 items are rated by a clinician on the basis of the child's nonverbal behavior. Items scales are 1 to 5 for sleep, appetite, and speech and 1 to 7 for the remaining 14 items. Total scores are summed and range from 17 to 113, with lower scores indicating normality while higher scores indicate psychopathology. Lower scores post-intervention indicate treatment efficacy.
  score | 55.9 (10.4) | 55.3 (11) | 55.6 (10.5)
Children's Global Assessment Scale [Mean (Standard Deviation); unit: score] — The Children's Global Assessment Scale (CGAS) is a numeric scale used by mental health clinicians to rate the general functioning. Scores range from 1 to 100, with high scores indicating better functioning. A score of 1-10 indicates the need for constant supervision, while a score of 91-100 indicates superior functioning.
  score | 50.4 (5.2) | 51.6 (6.9) | 51.0 (6.1)
Social Adjustment Scale-Self Report (SAS-SR) [Mean (Standard Deviation); unit: score] — The SAS-SR provides an understanding of an individual's level of satisfaction with his or her social situation, measuring the level of both behavioral and emotional social adjustment across four major areas (school, friends, family, and dating). Participants answer each item on a scale of 1 to 5. The total score also ranges from 1 to 5 and is the average of all item scores. The total score provides an index of social impairment with higher mean score indicating more difficulties with social adjustment. Lower scores post treatment indicate efficacy of the intervention.
  score | 2.8 (0.6) | 2.7 (.7) | 2.7 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: CDRS-R Score
Description: The CDRS-R is a clinician-administered semi-structured interview that assesses symptoms of depression experienced during the previous 2-weeks. The first 14 items are rated on the basis of an interview. The remaining 3 items are rated by a clinician on the basis of the child's nonverbal behavior. Items scales are 1 to 5 for sleep, appetite, and speech and 1 to 7 for the remaining 14 items. Total scores are summed and range from 17 to 113, with lower scores indicating normality while higher scores indicate psychopathology. Lower scores post-intervention indicate treatment efficacy.
Time Frame: Baseline and 16-weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point
Number analyzed (Participants) | 20 | 20
score on a scale | 34.94 (2.05) | 40.65 (2.05)

2. Primary Outcome: CGAS Score
Description: The Children's Global Assessment Scale (CGAS) is a numeric scale used by mental health clinicians to rate the general functioning. Scores range from 1 to 100, with high scores indicating better functioning. A score of 1-10 indicates the need for constant supervision, while a score of 91-100 indicates superior functioning.
Time Frame: Baseline and 16-weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point
Number analyzed (Participants) | 20 | 20
score on a scale | 66.52 (2.39) | 60.66 (2.39)

3. Primary Outcome: SAS-SR Score
Description: The SAS-SR provides an understanding of an individual's level of satisfaction with his or her social situation, measuring the level of both behavioral and emotional social adjustment across four major areas (school, friends, family, and dating). Participants answer each item on a scale of 1 to 5. The total score also ranges from 1 to 5 and is the average of all item scores. The total score provides an index of social impairment with higher mean score indicating more difficulties with social adjustment. Lower scores post treatment indicate efficacy of the intervention.
Time Frame: Baseline and 16-weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point
Number analyzed (Participants) | 20 | 20
score on a scale | 2.16 (0.13) | 2.35 (0.14)

ADVERSE EVENTS:
Time Frame: 16-weeks
Arm/Group | Talk Therapy 4-Week Decision Point | Talk Therapy 8-Week Decision Point
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/20
Other Adverse Events (participants affected / at risk) | 11/20 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talk Therapy 4-Week Decision Point (N=20) | Talk Therapy 8-Week Decision Point (N=20)
Suicide Attempt (Psychiatric disorders) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talk Therapy 4-Week Decision Point (N=20) | Talk Therapy 8-Week Decision Point (N=20)
Harm-related (Psychiatric disorders) | 6 | 8
Suicide-Related (Psychiatric disorders) | 5 | 4 — A suicide-related adverse event was defined as worsening suicidal ideation, a suicide attempt, or both.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No